CLINICAL TRIAL: NCT00981617
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled, Adaptive Study of the Safety and Efficacy of RDC-0313 in Adults With Alcohol Dependence
Brief Title: ALK33-005: A Study of ALKS33 (RDC-0313) in Adults With Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK33-005
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — ALKS-33

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ALKS33 (RDC-0313) (1 mg) (Experimental): 1 mg ALKS33 (RDC-0313) provided as capsules for daily oral administration
  Interventions: Drug: ALKS33 (RDC-0313) (1 mg)
- ALKS33 (RDC-0313) (2.5 mg) (Experimental): 2.5 mg ALKS33 (RDC-0313) provided as capsules for daily oral administration
  Interventions: Drug: ALKS33 (RDC-0313) (2.5 mg)
- ALKS33 (RDC-0313) (10 mg) (Experimental): 10 mg ALKS33 (RDC-0313) provided as capsules for daily oral administration
  Interventions: Drug: ALKS33 (RDC-0313) (10 mg)
- Placebo (Placebo Comparator): Matching placebo (capsules without active study drug) provided for daily oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS33 (RDC-0313) (1 mg) — 1 mg ALKS33 (RDC-0313) taken once daily for 12 weeks
  Arms: ALKS33 (RDC-0313) (1 mg)
Drug: ALKS33 (RDC-0313) (2.5 mg) — 2.5 mg ALKS33 (RDC-0313) taken once daily for 12 weeks
  Arms: ALKS33 (RDC-0313) (2.5 mg)
Drug: ALKS33 (RDC-0313) (10 mg) — 10 mg ALKS33 (RDC-0313) taken once daily for 12 weeks
  Arms: ALKS33 (RDC-0313) (10 mg)
Drug: Placebo — Matching placebo taken once daily for 12 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of ALKS33 (RDC-0313) compared with placebo in adults with alcohol dependence. There will be 11 study visits conducted over a period of about 4 months. The study period includes a screening visit, a 12-week treatment period, and a follow-up visit.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study. A 3-stage adaptive design will be used. Following screening, eligible subjects will be randomized equally to 1 of 4 groups (ALKS33 [RDC-0313] [1, 2.5, OR 10 mg], or matching placebo).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current diagnosis of alcohol dependence, with recent heavy drinking (eg, 5 drinks per day for men and 4 drinks per day for women)
* A noncustodial stable residence and a telephone
* Women having reproductive potential must agree to use an approved method of contraception for the duration of the study
* Ability to stop drinking prior to receiving study drug

Exclusion Criteria:

* Pregnancy and/or current breastfeeding
* Past or present history of an AIDS-indicator disease
* Current dependence on any drugs (exclusive of nicotine, caffeine, or alcohol)
* Positive urine drug screen for benzodiazepines (unless used for a short-term basis during alcohol detoxification), opioids, amphetamines/ methamphetamines or cocaine at Visits 1 and 2
* Clinically significant medical condition
* Current or anticipated need for prescribed opioid medication during the study period
* Use of naltrexone within 60 days prior to screening
* Current need for antidepressants (within 30 days prior to entry)
* Participation in a clinical trial of a pharmacological agent within 30 days prior to screening
* Parole or probation or pending legal proceedings that have the potential for incarceration during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Percent of subjects abstinent from heavy drinking | 12 Weeks

SECONDARY OUTCOMES:
Percent of subjects abstinent from any drinking | 12 Weeks
Percent of days abstinent from heavy drinking | 12 Weeks
Percent of days abstinent from any alcohol | 12 Weeks
Number of drinks per drinking day | 12 Weeks
Days to relapse to first heavy drinking day | 12 Weeks
Incidence of Adverse Events | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Cerritos, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Jacksonville, Florida
  - Alkermes Investigational Site, Maitland, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes Investigational Site, South Miami, Florida
  - Alkermes Investigational Site, West Palm Beach, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Roswell, Georgia
  - Alkermes Investigational Site, Lafayette, Indiana
  - Alkermes Investigational Site, Fall River, Massachusetts
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Albuquerque, New Mexico
  - Alkermes Investigational Site, Brooklyn, New York
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, Charlotte, North Carolina
  - Alkermes Investigational site, Hickory, North Carolina
  - Alkermes Investigational Site, New Bern, North Carolina
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Salt Lake City, Utah
  - Alkermes Investigational Site, Middleton, Wisconsin

REFERENCES:
- [Derived] O'Malley SS, Todtenkopf MS, Du Y, Ehrich E, Silverman BL. Effects of the Opioid System Modulator, Samidorphan, on Measures of Alcohol Consumption and Patient-Reported Outcomes in Adults with Alcohol Dependence. Alcohol Clin Exp Res. 2018 Oct;42(10):2011-2021. doi: 10.1111/acer.13849. Epub 2018 Aug 13. PMID 30055046